CLINICAL TRIAL: NCT05476185
Title: U.S. Committee for Refugees and Immigrants' READY4Life Program
Brief Title: USCRI READY4Life Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: US Committee for Refugees and Immigrants (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Young, Principal Investigator, US Committee for Refugees and Immigrants
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-06-29; First posted 2022-07-27 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Communication; Problem Solving; Social Relationships; Economic Stability
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned, in a three to one ratio, to the intervention group, or the control group. All participants will complete a pretest questionnaire and have access to case management services. The intervention group will receive 16 hours of Relationship Enhancement Education, then all participants will complete a posttest questionnaire. Six months after the posttest, all participants will complete a follow-up questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- READY4Life Programming - classroom instruction (Experimental): The intervention is an 16-hour classroom-based relationship education program taught by project staff. This instruction will strengthen and promote healthy marriages among young refugees and immigrants through education and comprehensive case management that will support an overall goal of helping youth build healthy relationship skills while supporting positive socio-emotional development and promoting successful transitions to young adulthood.
  Interventions: Behavioral: READY4Life Programming - classroom instruction
- No Intervention: Control (No Intervention): The control group does not receive any part of the classroom instruction that the intervention group receives. Like the intervention group, however, the control group does have access to case management.

INTERVENTIONS:
Behavioral: READY4Life Programming - classroom instruction — The intervention group receives 16 hours of classroom instruction.
  Arms: READY4Life Programming - classroom instruction

SUMMARY:
The U.S. Committee for Refugees and Immigrants (USCRI) has developed the Relationships, Education, Advancement, and Development for Youth for Life (READY4Life) Program. This is a 16-hour program for immigrants/refugees, ages 14 to 24. The program is designed to help young immigrants and refugees prepare for a successful life in the United States. The program is taught by USCRI program staff and is being implemented at eight sites across the U.S.: Cleveland, Ohio; Colchester, Vermont; Des Moines, Iowa; Miami, Florida; Philadelphia, Pennsylvania; Raleigh, North Carolina; Saint Paul, Minnesota; and Twin Falls, Idaho. The project also includes a rigorous evaluation component, featuring a Randomized Control Trial (RCT) design.

DETAILED DESCRIPTION:
The U.S. Committee for Refugees and Immigrants (USCRI) has developed the Relationships, Education, Advancement, and Development for Youth for Life (READY4Life) Program. This is a 16-hour program for immigrants/refugees, ages 14 to 24. The program is designed to help young immigrants and refugees prepare for a successful life in the United States. The program is taught by USCRI program staff and is being implemented at eight sites across the U.S.: Cleveland, Ohio; Colchester, Vermont; Des Moines, Iowa; Miami, Florida; Philadelphia, Pennsylvania; Raleigh, North Carolina; Saint Paul, Minnesota; and Twin Falls, Idaho. The project also includes a rigorous evaluation component, featuring a Randomized Control Trial (RCT) design.

Relationships, Education, Advancement, and Development for Youth for Life (READY4Life) will strengthen and promote healthy marriages among young refugees and immigrants through education and comprehensive case management that will support an overall goal of helping youth build healthy relationship skills while supporting positive socioemotional development and promoting successful transitions to young adulthood. USCRI's READY4Life program will serve refugee and immigrant youth ages 14 to 24, including but not limited to those individuals receiving, or who previously received TANF and/or individuals who are eligible for TANF assistance; non-custodial and custodial single parents; low-income, at-risk individuals; parenting youth; individuals with disabilities; and other eligible demographics, with a focus on underserved populations.

The Relationship Education curriculum, that was successfully used with an adult refugee/immigrant population, has been adapted for youth into a 16-hour curriculum composed of 1-, 2- and 4-hour sessions. Sessions are spaced a week apart to accommodate both federal requirements and research that shows relationship skills are best learned when practiced over time. . READY4Life will include ten communication and conflict resolution skills, as well as content information about effects of trauma on emotional stability and relationships, characteristics and advantages of healthy marriage, setting and achieving financial priorities and goals. Adaptations of the four core skills are taught: Expression Skills, Showing Understanding Skills, Discussion Skills, and Problem-Solving Skills. In the remaining hours of the curriculum, six additional skills are taught: Coaching and Conflict Management Skills, Self-Change and Helping Others Change Skills, and Generalization Skills and Maintenance Skills. Though not a part of the 10 Relationship Enhancement skills, time will also be devoted to financial management and making progress towards greater economic stability.

The four primary research questions deal with: 1) Communication skills; 2) Conflict resolution, conflict management, and problem-solving skills; 3) Healthy relationship and marriage skills; 4) Progress towards greater economic stability. We have selected these research questions because we believe, and the literature supports the position, that these factors are of major importance in helping youth make a successful transition from adolescence to adulthood.

The intervention participants will receive the IDEALS curriculum for community participants ages 14 to 24. Total: 16 hours per intervention participant (3,600 total intervention participants).

The control group will not receive the curriculum (1,200 total control participants). Note: once the control participants have completed the pre-test questionnaire, post-test questionnaire and six-month follow-up, they will be eligible to receive the intervention services, but they will not be counted as an intervention participant. Their participation in the evaluation will end once the six-month follow-up questionnaire is collected.

Educational Evaluators, Inc. (EEI) is the local evaluator on this project working with USCRI's READY4Life Program. We also want grantee staff to understand the importance of evaluation and to be familiar with the evaluation protocols. By working closely together from the initial development of the proposal and picking up that collaboration as soon as the grant award was made, the evaluation staff and the grantee staff work together to understand all dimensions of the program. We believe this strengthens the overall evaluation, since EEI is not simply looking in as outsiders, but has provided training in all evaluation procedures to all grantee project staff including the Project Director, Program Coordinators, and Data Collection Specialists. This again, strengthens the evaluation.

Random Assignment. Participants will be randomly assigned the intervention group or the control group in a 3:1 ratio. Thus, of the total number of participants per year, 25% will be assigned to the control group, and the remaining 75% will be assigned to the intervention group. The evaluation team will use a random number generator created by Qualtrics to assign subjects to the intervention or control as described above. Demographic data for the intervention group will be compared with the control group to determine whether there are group differences on any of the demographic variables. If differences are detected between an intervention group and control group, then that variable will be used as a co-variate when comparing groups relative to outcome variables.

The unit of analysis will be the individual participant, refugee/immigrant youth, ages 14-24. Many participants will be youth enrolled in high school grades 9-12, although participants up to the age of 24 will be eligible for enrollment. The program will not be provided during the school day, as part of the school curriculum. Some schools, however, will allow us to use the school facilities to provide the program in an after-school setting. The schools providing after-school settings have high percentages of English Language Learners and immigrant and refugee student populations. Several are part of the Refugee School Impact Working Group, offer the Success Management Academy Program targeting recent arrivals to the US, or come from districts offering Newcomer Centers serving immigrant and refugee students.

This project targets low-income and at-risk, refugee and immigrant youth, ages 14-24. The target population will not differ from those who will be broadly served by the grant. Participants will be young people who self-identify as refugees or immigrants.

An instrument was developed after a comprehensive review of the intervention to be implemented. This instrument is aligned with the research questions and hypotheses developed. The Local Evaluation Questionnaire (LEQ) contains 5 demographic questions and 55 questions to answer the primary and secondary research questionsThe four primary research questions deal with: 1) Communication skills; 2) Conflict resolution, conflict management, and problem-solving skills; 3) Healthy relationship and marriage skills; 4) Progress towards greater economic stability. We have selected these research questions because we believe, and the literature supports the position, that these factors are of major importance in helping youth make a successful transition from adolescence to adulthood.

Statistical Power. Statistical power for evaluation of this study's hypotheses was calculated using Optimal Design Software for Multilevel and Longitudinal Research Version 3.01. Power calculations were computed to estimate minimum detectable effect sizes based on group comparisons over time, with an alpha of .05 and power of .80.

Adequate power to detect small to moderate effect sizes (δ = .35) will be present if the total variance in the outcomes explained by the difference between groups is small (intervention correlation ρ =.05). If the intervention correlation is moderate (ρ = 0.10), the minimum detectable effect size will be moderate (δ = 0.46). With a much smaller sample, Denny and Young (2006) found statistically significant results for changes in knowledge, attitudes, hopelessness, self-efficacy, and sexual intent, with effect sizes, measured by Eta square, ranging from .029-.170. Based on this previous work, we feel confident the study will be sufficiently powered to examine the effects of interest.

Statistical Analyses. Frequency counts and percentages will be used to report the characteristics of the sample. Factor analysis will be used to confirm that the items comprising a given variable load together on a single factor. Cronbach's alpha will be used to examine internal consistency of the items comprising the four outcome variables. Descriptive statistics will be used, reporting means and standard deviations for the four outcome variables. Differences by group, relative to demographic variables, such as gender and race, will be examined using chi-square. Data will also be analyzed using analysis of covariance. The pretest score of the outcome measure under consideration will be used as the covariate. Data will again be analyzed using analysis of covariance, but not only using the pretest score as a covariate, but also treatment dose level, and nationality.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 14 years old and no more than 24 years old
* Must self-identify as a refugee or immigrant

Exclusion Criteria:

* Younger than 14 years old or older than 24 years old
* Does not identify as a refugee or immigrant

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4800 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Healthy Communication Skills Score | Time Frame: Pretest to Follow-up (six months after completion of the intervention - about 7 months after the pretest)
  This outcome is the participants' score on a healthy marriage/relationship skills scale. This is a 10 item scale. It was used in an article recently published in Family Relations. The principal investigator for the present study (Young) was also the lead author for the study published in Family Relations. A sample item from the scale is "It is important to show appreciation for others." In the Family Relations study the items in the scale loaded on a single factor at .56 or above. The internal consistency (Chronbach's alpha) at pretest was .87. The percentage of the variance explained by the first component was 46. The results table will report the mean scores of the intervention and control groups at pretest, posttest and follow-up, as well as the results from the statistical analysis.
Conflict Resolution, Management, and Problem-Solving Skills Score | Time Frame: Pretest to Follow-up (six months after completion of the intervention - about 7 months after the pretest)
  This outcome is the participants' score on a conflict management/ resolution skills scale. This is a 6 item scale. It was used in an article recently published in Family Relations. The principal investigator for the present study (Young) was also the lead author for the study published in Family Relations. A sample item from the scale is "I follow through on promises and agreements." In the Family Relations study the items in the scale loaded on a single factor at .60 or above. The internal consistency (Chronbach's alpha) at pretest was .83. The percentage of the variance explained by the first component was 54.The results table will report the mean scores of the intervention and control groups at pretest, posttest and follow-up, as well as the results from the statistical analysis.
Healthy Relationship and Marriage Skills Score | Time Frame: Pretest to Follow-up (six months after completion of the intervention - about 7 months after the pretest)
  This outcome is the participants' score on a healthy relationship and marriage skills scale. This is a 6 item scale. A sample item from the scale is "In times of crisis we can turn to each other for support." The results table will report the mean scores of the intervention and control groups at pretest, posttest and follow-up, as well as the results from the statistical analysis.
Progress Toward Greater Economic Stability | Time Frame: Pretest to Follow-up (six months after completion of the intervention - about 7 months after the pretest)
  This outcome is the participants' score on an attitudes about personal finances scale. This is a 6 item scale. It was used in an article recently published in Family Relations. The principal investigator for the present study (Young) was also the lead author for the study published in Family Relations. A sample item from the scale is "I can reduce conflict about money through discussion and problem solving." In the Family Relations study the items in the scale loaded on a single factor at .63 or above. The internal consistency (Chronbach's alpha) at pretest was .72 and .94 at posttest.The results table will report the mean scores of the intervention and control groups at pretest, posttest and follow-up, as well as the results from the statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Young, Ph.D., Principal Investigator — Educational Evaluators, Inc; Center for Evidence-Based Programming
Locations (9):
- United States (9):
  - United States Committe on Refugees and Immigrants, Washington D.C., District of Columbia
  - Youth Coop Inc., Miami, Florida
  - College of Southern Idaho Refugee Program, Twin Falls, Idaho
  - USCRI Des Moines, Des Moines, Iowa
  - Internationa Institute of Minnesota, Saint Paul, Minnesota
  - USCRI North Carolina, Raleigh, North Carolina
  - USCRI Cleveland, Cleveland, Ohio
  - Nationalities Service Center, Philadelphia, Pennsylvania
  - USCRI Vermont, Colchester, Vermont